CLINICAL TRIAL: NCT00736047
Title: A Double Blind, Placebo-controlled, Multi-centre Study to Evaluate the Efficacy, Safety, Tolerability and Immunogenicity of Repeated s.c Administrations of 100µg NIC002 Vaccine in Cigarette Smokers Who Are Motivated to Quit Smoking.
Brief Title: Study to Evaluate the Efficacy, Safety, Tolerability and Immunogenicity of 100µg NIC002 Vaccine in Cigarette Smokers Who Are Motivated to Quit Smoking.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNIC002A2201
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Smokers
Keywords: Smokers; smoking cessation; vaccine; antibodies; anti-nicotine
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Biological: NIC002
- 2 (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NIC002
  Arms: 1
Biological: Placebo
  Arms: 2

SUMMARY:
This study is designed to determine the efficacy of high nicotine-specific antibody titers in smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female smoking subjects age 18 to 65 years of age
* Subjects must be smoking 10 or more cigarettes per day during the past 12 months
* The exhaled breath carbon monoxide (CO) concentration must be 10 ppm or more at screening. Urine cotinine at screening must be positive.
* The Fagerström Test for Nicotine Dependence (FTND) score of 5 or above at screening.

Exclusion Criteria:

* Attempted to quit smoking in the three (3) months.
* Prior use of smoking cessation aid.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Smoking status | 12 weeks
Exhaled carbon monoxide | 12 weeks

SECONDARY OUTCOMES:
Smoking status at various time intervals from target quit date to the end of the study | 52 weeks
Safety and tolerability | 52 weeks
Immunogenicity (specific anti-nicotine antibodies in serum) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis Investigator Site
Locations (2):
- Germany (2):
  - Novartis Investigative Site, Mainz
  - Novartis Investigator Site, Neuss